CLINICAL TRIAL: NCT05041270
Title: Epidural Nalbuphine Versus Dexmedetomidine as Adjuvants to Bupivacaine in Lower Limb Surgeries Under Combined Spinal-epidural Anesthesia
Brief Title: Epidural Nalbuphine Versus Dexmedetomidine as Adjuvants to Bupivacaine in Lower Limb Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Rehab Abd-Allah Wahdan, lecturer of anesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-8-2021
Record Dates: First submitted 2021-09-02; First posted 2021-09-13 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Lower Limb Surgeries
Keywords: Epidural Nalbuphine; Epidural Dexmedetomidine; combined spinal-epidural anesthesia; lower limb surgeries
MeSH Terms: interventions — Saline Solution; Dexmedetomidine; Nalbuphine

STUDY DESIGN:
Intervention Model Description: The patients will be divided randomly by a computer-generated randomization table into three equal groups
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: triple blinded (patient, anesthesiologist in the operating room and outcomes assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Placebo Comparator): patient will be given epidural bolus dose of 12ml (10ml 0.25% bupivacaine + 2ml normal saline), top up dose of 8ml will be given postoperative (6ml 0.25% bupivacaine + 2ml normal saline).
  Interventions: Drug: normal saline
- dexmedetomidine group (Active Comparator): patient will be given epidural bolus dose of 12ml (10ml 0.25% bupivacaine + 100µg dexmedetomidine in 2ml volume), top up dose of 8ml will be given postoperative (6ml 0.25% bupivacaine + 20µg dexmedetomidine in 2ml volume)
  Interventions: Drug: Dexmedetomidine
- nalbuphine group (Active Comparator): patient will be given epidural bolus dose of 12ml (10ml 0.25% bupivacaine + 10mg nalbuphine in 2ml volume), top up dose of 8ml will be given postoperative (6ml 0.25% bupivacaine + 2mg nalbuphine in 2ml volume)
  Interventions: Drug: Nalbuphine

INTERVENTIONS:
Drug: normal saline — Surgery will be started under spinal anesthesia. When sensory block regress to T12 dermatome Epidural bolus dose will be given epidural bolus dose of 12ml (10ml 0.25% bupivacaine + 2ml normal saline) The onset of sensory blockade injected epiduraly with maximal cephalic spread will be assessed by bilateral pinprick method along the midclavicular line, every 5 min for 30 min and then every 30 min.
  top up dose of 8ml will be given postoperative (6ml 0.25% bupivacaine + 2ml normal saline).
  Arms: control group
Drug: Dexmedetomidine — Surgery will be started under spinal anesthesia. When sensory block regress to T12 dermatome Epidural bolus dose will be given epidural bolus dose of 12ml (10ml 0.25% bupivacaine + 100µg dexmedetomidine in 2ml volume) The onset of sensory blockade injected epiduraly with maximal cephalic spread will be assessed by bilateral pinprick method along the midclavicular line, every 5 min for 30 min and then every 30 min.
  top up dose of 8ml will be given postoperative (6ml 0.25% bupivacaine + 20µg dexmedetomidine in 2ml volume).
  Arms: dexmedetomidine group
Drug: Nalbuphine — Surgery will be started under spinal anesthesia. When sensory block regress to T12 dermatome Epidural bolus dose will be given epidural bolus dose of 12ml (10ml 0.25% bupivacaine + 10mg nalbuphine in 2ml volume) The onset of sensory blockade injected epiduraly with maximal cephalic spread will be assessed by bilateral pinprick method along the midclavicular line, every 5 min for 30 min and then every 30 min.
  top up dose of 8ml will be given postoperative (6ml 0.25% bupivacaine + 2mg nalbuphine in 2ml volume).
  Arms: nalbuphine group

SUMMARY:
Combined spinal epidural anesthesia (CSE) with bupivacaine alone is not sufficient to cover pain sequel during lower limb surgeries.

Previous studies used addition of either Nalbuphine or dexmedetomidine to bupivacaine in epidural anesthesia giving a good result in pain control.

In this study the investigators will evaluate and compare the addition of either Nalbuphine or dexmedetomidine to bupivacaine in epidural anesthesia to evaluate the analgesic efficacy of either drug.

DETAILED DESCRIPTION:
Surgical patients need adequate and effective intraoperative anesthesia and postoperative analgesia. Neuroaxial block including lower limb spinal and epidural blocks have a long history of effective anesthesia and lower limb pain relief. Spinal anesthesia is a simple method requiring small dose of local anesthetic agent to give immediate and effective sensory and motor block. But one of its major side effects is hypotension and difficulty in controlling the level of the block [1]. Meanwhile, epidural anesthesia is a safe, well-practiced, not expensive neuroaxial block technique that provides intraoperative anesthesia and postoperative analgesia. So, the combined spinal epidural block (CSE) aims to achieve intense sensory and motor anesthesia and prolong the duration of analgesia intraoperative extending to postoperative period [2].

Neuroaxial anesthesia and analgesia provide perfect analgesic effect by inhibiting nociceptive transmission from peripheral to central neuronal system, but this advantage limited by short half-life of the current local anesthetics. Bupivacaine is a local anesthetic which belongs to amide group of anesthetic agents that has been widely used for local infiltration, peripheral nerve block, spinal and epidural anesthesia and despite relatively long duration of action, still has insufficient time for postoperative analgesia [3].

Several neuroaxial adjuvants such as (opioids, dexamethasone, magnesium sulphate, midazolam and dexmedetomidine) can be added to local anesthetics to prolong its duration of anesthesia and decrease the dose requirement of local anesthetics [4].

Nalbuphine, a derivative of 14-hydroxy morphine is a strong analgesic with mixed kappa agonist and µ antagonist properties. Its potency is equal to morphine, but exhibits a ceiling effect on respiratory depression. It has the potential to maintain and enhance µ-opioid based anesthesia while simultaneously mitigating the µ-opioid side effects [5].

Dexmedetomidine is an imidazole compound. It is a highly selective α-2 adrenergic agonist with an affinity 8 times more specific when compared to clonidine. It has sedative, sympatholytic and analgesic effects that blunt cardiovascular responses both intraoperative and in the perioperative period. Patients remain calm and sedated when undisturbed but arouse readily with stimulation [6]. Dexmedetomidine causes manageable hypotension and bradycardia, but the striking feature of this drug is the lack of opioid-related adverse effects like respiratory depression, pruritis, nausea, and vomiting [7].

ELIGIBILITY:
Inclusion Criteria:

* patient acceptance.
* BMI 25-29.9 kg/m2.
* ASA I and ASA II.
* Scheduled for elective lower limb orthopedic surgeries under (CSE) block.

Exclusion Criteria:

* Patient with known allergy to study drugs,
* Patients suffering from severe chronic diseases (cardiac, renal, hepatic and neurological or diabetes),
* Patients with infection at the site of spinal-epidural block,
* Drug addict patients,
* Patients on long term steroid therapy,
* Patients with abnormalities in vertebral spine,
* Mentally retarded or uncooperative patients,
* Patients receive anti-coagulant therapy or suspected coagulopathy.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Duration of epidural analgesia | within 24 hour postoperative
  time elapsed from epidural injection of LA until VAS score (≥3)
Maximum level of sensory blockade | after 30 min of administering the local anesthetic in the epidural space
  the maximum sensory dermatome level after 30 min of administering the local anesthetic in the epidural space

SECONDARY OUTCOMES:
number of top up doses required | within 24 hour postoperative
  When sensory block regress to T12 dermatome Epidural bolus dose will be given
assessment of changes in patient's level of sedation | Sedation scores will be recorded just before the initiation and 2 hours postoperatively
  assessment of patient's level of sedation using Ramsey sedation score; where 1=patient is anxious and agitated or restless, or both.
  2= Patient is co-operative, oriented, and tranquil. 3= Patient responds to commands only. 4= Patient exhibits brisk response to light glabellar tap or loud auditory stimulus.
  5= Patient exhibits a sluggish response to light glabellar tap or loud auditory stimulus.
  6= Patient exhibits no response.

CONTACTS AND LOCATIONS:
Overall Officials: Howaida A Kamal, MD, Study Director — Faculty of medicine, zagazig university, Zagazig, Elsharqya, Egypt, 44519
Locations (1):
- faculty of medicine, Zagazig university, Zagazig, Elsharqya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planned after the completion of the study and publication
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: planned after the completion of the study and publication
Access Criteria: principal investigator

REFERENCES:
- [Background] Shruthi AH, Sudheesh K, Nethra SS, Raghavendra Rao RS, Devika Rani D. THE EFFECT OF A SINGLE DOSE OF MAGNESIUM SULPHATE AS AN ADJUVANT TO EPIDURAL BUPIVACAINE FOR INFRAUMBILICAL SURGERIES: A PROSPECTIVE DOUBLE-BLIND, RANDOMIZED CONTROL TRIAL. Middle East J Anaesthesiol. 2016 Feb;23(4):449-55. PMID 27382815
- [Background] Chatrath V, Attri JP, Bala A, Khetarpal R, Ahuja D, Kaur S. Epidural nalbuphine for postoperative analgesia in orthopedic surgery. Anesth Essays Res. 2015 Sep-Dec;9(3):326-30. doi: 10.4103/0259-1162.158004. PMID 26712968
- [Background] Gupta K, Rastogi B, Gupta PK, Singh I, Bansal M, Tyagi V. Intrathecal nalbuphine versus intrathecal fentanyl as adjuvant to 0.5% hyperbaric bupivacaine for orthopedic surgery of lower limbs under subarachnoid block: A comparative evaluation. Indian J Pain. 2016; 30:90-5.
- [Background] Chiruvella S, Donthu B, Nallam SR, Salla DB. Postoperative Analgesia with Epidural Dexmedetomidine Compared with Clonidine following Total Abdominal Hysterectomies: A Prospective Double-blind Randomized Trial. Anesth Essays Res. 2018 Jan-Mar;12(1):103-108. doi: 10.4103/aer.AER_207_17. PMID 29628563
- [Background] Soliman AAM, Melika ASM. Epidural bupivacaine and dexmedetomidine versus bupivacaine and opioids for lower vascular surgery. J Med Sci Res. 2018; 1:158-63.
- [Background] Paul A, Nathroy A, Paul T. A comparative study of dexmedetomidine and fentanyl as an adjuvant to epidural bupivacaine in lower limb surgeries. J Med Sci. 2017; 37:221-6.
- [Derived] Farmawy MSE, Mowafy SMS, Wahdan RA. Epidural nalbuphine versus dexmedetomidine as adjuvants to bupivacaine in lower limb orthopedic surgeries for postoperative analgesia: a randomized controlled trial. BMC Anesthesiol. 2023 Dec 6;23(1):401. doi: 10.1186/s12871-023-02348-x. PMID 38057695